CLINICAL TRIAL: NCT02803671
Title: Analysis of the Impact of Patent Ductus Arteriosus on Brain Function in Preterm Neonates: Multimodal Approach Integrating EEG-NIRS, Ultrasound and Clinical Data
Acronym: NNP-MULTIMODAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PHRCN08-DR-KONGOLO
Record Dates: First submitted 2016-06-10; First posted 2016-06-17 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Ductus Arteriosus, Patent
Keywords: preterm neonates; EEG-NIRS
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — Electroencephalography

ARMS (3):
- patent ductus arteriosus (Experimental): ultrasounds Transfontanellaires near-infrared spectroscopy (TFU-NIRS) near-infrared spectroscopy (NIRS) electroencephalogram (EEG)
  Interventions: Device: TFU-NIRS; Device: NIRS; Device: EEG
- without patent ductus arteriosus (Experimental): ultrasounds Transfontanellaires near-infrared spectroscopy (TFU-NIRS) near-infrared spectroscopy (NIRS) electroencephalogram (EEG)
  Interventions: Device: TFU-NIRS; Device: NIRS; Device: EEG
- patent ductus arteriosus + cardiac or respiratory therapy (Experimental): ultrasounds Transfontanellaires near-infrared spectroscopy (TFU-NIRS) near-infrared spectroscopy (NIRS) electroencephalogram (EEG)
  Interventions: Device: TFU-NIRS; Device: NIRS; Device: EEG

INTERVENTIONS:
Device: TFU-NIRS
Device: NIRS
Device: EEG

SUMMARY:
This project corresponds to the main field of research of the investigators's laboratory concerning analysis of cerebral electrometabolic and haemodynamic activity in neonates. In this context, the investigators have developed know-how and specific acquisition and analysis tools (2 patents and several publications), allowing them to apply this know-how in children with patent ductus arteriosus.

Patent ductus arteriosus after birth is characterized by shunting of a variable proportion of cardiac output towards the pulmonary circulation. The direct consequences of this shunting are: (i) overload of the pulmonary vasculature and left heart chambers, increasing the risk of left heart failure, haemorrhagic pulmonary oedema and late respiratory complications such as bronchopulmonary dysplasia; (ii) in contrast with the pulmonary circulation, other systemic organs are deprived of part of their normal perfusion and are subject to ischaemic hypoxia; the resulting neuronal hypoxia rapidly leads to metabolic and electrical dysfunction, the analysis of which constitutes one of the objectives of this project.

ELIGIBILITY:
Inclusion Criteria:

1. Group of children :

   * meeting the age criteria
   * having a ductus arteriosus persistence.
2. Group of children :

   * meeting the age criteria
   * with persistent ductus arteriosus in the ultrasound examination
   * for which a cardiac or respiratory treatment has already been put in place.
3. normal group of children :

   * meeting the age criteria
   * without ductus arteriosus persistence ultrasound or detectable neurological disorders after clinical, neurophysiological and radiological (ETF , Scanner, MRI).

Exclusion Criteria:

-

Max Age: 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2009-08-26 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
change in cerebral tissue oxygenation | Day 3, Day 5 , Day 12, week 5

CONTACTS AND LOCATIONS:
Overall Officials: Guy KONGOLO, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France